CLINICAL TRIAL: NCT02473861
Title: EXercise Influence on Taxane Side Effects (EXIT) Study
Acronym: EXIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: H15-00888
Record Dates: First submitted 2015-06-09; First posted 2015-06-17 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Breast Neoplasms
Keywords: exercise training; breast cancer; taxane chemotherapy; peripheral neuropathy; fatigue; autonomic function
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate exercise arm (Experimental): The length of the intervention for the immediate exercise group will be determined by treatment protocol and could range from 8 to 13 weeks. The intervention can begin up to one week before the first treatment and will continue until 2 weeks after the final taxane-containing treatment. The intervention will consist of thrice weekly supervised aerobic and resistance exercise training.
  Interventions: Other: Exercise
- delayed exercise arm (Experimental): The delayed exercise group will begin an exercise intervention two weeks after completion of their last taxane-containing chemotherapy treatment that will last the length of their taxane chemotherapy plus two weeks. If participants in the delayed exercise group have a surgery planned during the intervention time that will require >1 week off from exercise, the exercise intervention will be delayed until after the surgery. The intervention will consist of thrice weekly supervised aerobic and resistance exercise training.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Moderate intensity aerobic and resistance training. Five minutes each of warm-up, cool-down, balance and flexibility will also be performed.

SUMMARY:
This study is a randomized control cross over trial of exercise training during or after taxane-containing chemotherapy treatment for breast cancer. Forty-three women with stage I-III breast cancer will be randomized to immediate or delayed thrice weekly exercise training for 8-12 weeks. The immediate exercise group will exercise during taxane chemotherapy and the delayed group will start exercise 2 weeks after completion of treatment. This design will allow for an assessment of the effects of exercise vs usual care during treatment, plus a comparison of the training response during vs. after chemotherapy.

DETAILED DESCRIPTION:
Purpose The purpose of this study is to evaluate the effects of aerobic and resistance exercise training relative to usual care during taxane-containing chemotherapy treatment for breast cancer.

Hypotheses

Relative to usual care, aerobic and resistance exercise training during taxane-containing chemotherapy treatment for breast cancer will:

1. mitigate the experience of patient reported outcomes
2. reduce medical management of taxane side effects and adverse events
3. attenuate autonomic dysfunction and maintain resting cardiovascular function and cardiovascular response to exercise

4) Objectives The primary aim of this study is to determine whether aerobic and resistance exercise training during taxane-containing chemotherapy treatment reduces patient-reported side effects, medical management and clinical adverse events reported relative to usual care. The secondary aim is to determine the whether aerobic and resistance exercise training during taxane-containing chemotherapy attenuates the occurrence of indices of autonomic dysfunction relative to usual care.

5) Research methods This study is a randomized control trial with crossover. The intervention consists of aerobic, resistance and balance training three times a week. Forty-three women with a stage I-III breast cancer diagnosis who are scheduled to receive taxane-containing chemotherapy will be randomized to immediate or delayed exercise (stratified by treatment protocol). Potential participants will be referred by oncologist referral, or will be self-referred by recruitment posters, social media or word of mouth.

6) Statistical analysis The primary outcome measure is the EORTC CIPN subscale of patient-reported symptoms related to neurotoxic chemotherapy. Secondary outcome measures include measures of autonomic dysfunction including heart rate and blood pressure variability, and medical management of taxane-related side effects, and clinical adverse events related to treatment.

The chemotherapy-induced peripheral neuropathy (CIPN) sub-scale of the EORTC Quality of life Questionnaire is used as the primary outcome measure to determine sample size. G*Power 3.0.10 was used to estimate sample size for independent t-tests between the two groups (at the 2-week post chemotherapy time point). At thirty-six participants, we will have 80% power to detect a medium (d=0.6) effect size in the EORTC CIPN-20 subscale at an alpha of 0.05 (one-tailed) . An additional 20% will be recruited to allow for dropout or non-adherence, making the final total sample size goal 43 participants.

Baseline characteristics and outcome measures of the two groups will be compared with independent t-tests. To assess the effect of the exercise intervention during treatment, independent t-tests will be used to compare the outcome measures at two weeks post completion of taxane chemotherapy if no difference exists between groups baseline measures. For the exercise group, all outcome measures at time point 2 will be compared to time point 3 using paired t-tests to assess maintenance over time. Independent t-tests will first be used to determine whether significant differences exists between groups for the three exploratory measure time points. If no differences exist, all data will be combined, and analyzed with a repeated measures analysis of variance to determine whether differences exist.

ELIGIBILITY:
Inclusion Criteria:

* Born female
* Age 19 or older
* Histologically confirmed stage I-IIIA breast cancer diagnosis
* Scheduled to receive neoadjuvant or adjuvant taxane-containing chemotherapy
* Willing and able to attend baseline assessment prior to first taxane-containing treatment
* Have reliable transportation to attend our exercise gym located near the Vancouver BCCA three times weekly for 8-13 weeks
* Be able to read and communicate in English
* Treating medical oncologist approval to participate

Exclusion Criteria:

* Receipt of further chemotherapy treatments after taxane-containing treatments
* Stage IV cancer
* Acute or uncontrolled health conditions including heart disease, respiratory disease (COPD or severe asthma)
* Diagnosis of diabetes at any time
* Personal history of neurological disorder
* Mobility issues that require a mobility aid or that prevent exercise on a bike, treadmill, or elliptical (includes orthopedic injury or arthritis that result in inability to exercise)
* Body mass index ≥40 kg/m2
* Previously received chemotherapy or thoracic radiation treatment

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Change with treatment and maintenance post treatment in patient-reported taxane-related symptoms via the EORTC CIPN subscale | 14-0 days pre taxane chemotherapy, 1-2 weeks after completion of half of planned taxane chemotherapy treatments, 2 weeks post completion of taxane chemotherapy, 10-15 weeks post completion of taxane chemotherapy
  European Organization for Research and Treatment of Cancer CIPN subscale

SECONDARY OUTCOMES:
Change with treatment and maintenance post treatment of heart rate variability | 14-0 days pre taxane chemotherapy, 2 weeks post completion of taxane chemotherapy, 10-15 weeks post completion taxane chemotherapy
  Electrocardiography will be used to assess heart rate variability during 10 minutes of supine rest
Change with treatment and maintenance post treatment of blood pressure variability | 14-0 days pre taxane chemotherapy, 1-2 weeks after completion of half of planned taxane chemotherapy treatments, 2 weeks post completion of taxane chemotherapy, 10-15 weeks post completion of taxane chemotherapy
  A Finometer will be used to assess blood pressure variability from supine to standing posture
Number of participants requiring medical management of taxane side effects | Will be extracted from medical records 0-6 months after completion of chemotherapy
  Prescription of medications, dose delays, dose reductions will be abstracted from cancer treatment records
Number of participants with clinical reporting of adverse events during taxane-chemotherapy treatment | Will be extracted from medical records 0-6 months after completion of chemotherapy
  Oncological treatment notes will be reviewed for clinical notation of adverese events during taxane treatment

OTHER OUTCOMES:
Change with treatment and maintenance post treatment of aerobic fitness via estimated peak oxygen consumption | 14-0 days pre taxane chemotherapy, 2 weeks post taxane chemotherapy, 10-15 weeks post taxane chemotherapy
  Peak oxygen consumption be estimated from incremental cycle ergometer test
Change with treatment and maintenance post treatment of lower body muscular strength via estimated 1-repetition maximum leg press | 14-0 days pre taxane chemotherapy, 2 weeks post taxane chemotherapy, 10-15 weeks post taxane chemotherapy
  Lower body strength be assessed by estimated 1 repetition maximum leg press
Change with treatment and maintenance post treatment of upper body muscular strength via handgrip strength | 14-0 days pre taxane chemotherapy, 2 weeks post taxane chemotherapy, 10-15 weeks post taxane chemotherapy
  Handgrip strength will be assessed via handgrip dynamomemeter
Change during treatment and post treatment in cancer-related fatigue via revised Piper Fatigue Scale | 14-0 days pre taxane chemotherapy, 0-3 days pre chemo cycle 3, 3-5 days post chemo cycle 3, 0-3 days pre chemo cycle 4, 2 weeks post taxane chemotherapy, 10-15 weeks post taxane chemotherapy
  Revised Piper Fatigue Scale will be administered electronically to assess change with the intervention but also across one cycle (third) of chemotherapy to investigate patterns in fatigue
Change in pain with treatment and improvement post treatment via Brief Pain Inventory | 14-0 days pre taxane chemotherapy, 2 weeks post taxane chemotherapy, 10-15 weeks post taxane chemotherapy
  The Brief Pain Inventory will be administered electronically

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Breast Cancer Training Center, 614 W. 8th Ave, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided